CLINICAL TRIAL: NCT00233181
Title: Adherence Intervention for Minority Children With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 298; R01HL052013 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Behavioral: Home-based adherence monitoring

SUMMARY:
To evaluate the effectiveness of a Head Start-based early intervention for designed to improve asthma management skill and practices of parents, pre-school children and Head Start staff.

DETAILED DESCRIPTION:
BACKGROUND:

While increased asthma morbidity and mortality have been observed across all ethnicities, results from several studies have found that asthma morbidity has increased disproportionately in low-income African American children. Elementary school-based asthma education programs have shown promise in improving asthma management, and reducing asthma morbidity in this high-risk population, however, the fastest growing asthma risk is associated with children young than six. By elementary age many parents and children with asthma have well-established patterns of inappropriate asthma management that may be difficult to change. To date, no research has examined the impact of early intervention for asthma management in low-income, high-risk children.

DESIGN NARRATIVE:

The primary outcome that the study was designed to evaluate medical record documented emergency care for asthma at the JHPED over the eighteen-month follow-up period.

The secondary outcomes Adherence with asthma therapy based on Medicaid pharmacy claims for asthma medications, other asthma health care (urgent and primary), self-reported medication adherence, barriers to health care, restricted activity, nighttime symptoms, asthma medications, self and family asthma management behaviors, asthma management self-efficacy, functional status, and quality of life.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
1. Age 2-12 years.
2. A current diagnosis of asthma or reactive airway disease
3. Resident of Baltimore City.
4. Two or more ED visits at the JHPED for asthma in the past 12 months, or hospitalization for asthma at the JHPED in the past 12 months by parent report.
5. Not currently participating in other research studies (participation in previous studies will be noted).

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2000-04; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Rand — Johns Hopkins University

REFERENCES:
- [Background] Paasche-Orlow MK, Riekert KA, Bilderback A, Chanmugam A, Hill P, Rand CS, Brancati FL, Krishnan JA. Tailored education may reduce health literacy disparities in asthma self-management. Am J Respir Crit Care Med. 2005 Oct 15;172(8):980-6. doi: 10.1164/rccm.200409-1291OC. Epub 2005 Aug 4. PMID 16081544
- [Derived] Otsuki M, Eakin MN, Rand CS, Butz AM, Hsu VD, Zuckerman IH, Ogborn J, Bilderback A, Riekert KA. Adherence feedback to improve asthma outcomes among inner-city children: a randomized trial. Pediatrics. 2009 Dec;124(6):1513-21. doi: 10.1542/peds.2008-2961. PMID 19948623